CLINICAL TRIAL: NCT04855422
Title: Assessing Benchmarks For Allosure And Allomap Testing in Simultaneous Kidney & Pancreas Transplant Recipients.
Acronym: SPKCareDx
Status: Active, not recruiting | Type: Observational
Sponsor: Montefiore Medical Center (Other)
Collaborators: CareDx (Industry)
Responsible Party: Sponsor
Other Study IDs: 2021-12823
Record Dates: First submitted 2021-04-19; First posted 2021-04-22 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Transplant; Complication, Rejection
MeSH Terms: conditions — Rejection, Psychology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Stable SPK recipients without rejection and/or BKV viremia: All SPK transplant recipients are monitored for routine labs twice a week first month, weekly at 2nd and 3rd month, every 2 weeks between 3-6 months, once a month between 6-12 months and then once every 2 months.
  Interventions: Diagnostic Test: Allosure; Diagnostic Test: AlloMap
- Acute T-Cell Mediated Rejection (TCMR ): Kidney and pancreas transplant biopsies will be solely for clinically indicated for increased creatinine, amylase, lipase, blood sugar levels of more than 20% of the baseline, increased spot urine protein/creatinine ratio more than 1 gram/day, and development of donor-specific anti-Human Leukocyte Antigen (anti-HLA) antibodies.
  Interventions: Diagnostic Test: Allosure; Diagnostic Test: AlloMap
- Antibody Medicated Rejection (ABMR): Kidney and pancreas transplant biopsies will be solely for clinically indicated for increased creatinine, amylase, lipase, blood sugar levels of more than 20% of the baseline, increased spot urine protein/creatinine ratio more than 1 gram/day, and development of donor-specific anti-HLA antibodies.
  Interventions: Diagnostic Test: Allosure; Diagnostic Test: AlloMap
- BKV viremia: All patients will be monitored for BKV viremia monthly after transplantation up to 6 months and at 9, 12 and 24 months. Luminex Single Antigen Bead (SAB) will be monitored at 1, 3, 12 and 24 months. Spot urine protein and creatinine and HbA1c will be monitored every 3 months after transplantation
  Interventions: Diagnostic Test: Allosure; Diagnostic Test: AlloMap
- Follow-up of subjects with acute TCMR, ABMR and BKV viremia after treatment: BKV viremia, Luminex SAB, spot urine protein and creatinine is studied at the time clinically indicated biopsy and/o worsening kidney function and proteinuria.
  Interventions: Diagnostic Test: Allosure; Diagnostic Test: AlloMap

INTERVENTIONS:
Diagnostic Test: Allosure — AlloSure Analysis For the AlloSure test, 10-20 mL of blood will be obtained in Streck Cell-Free DNA blood collection tubes (BCT) and shipped to CareDx, Inc. (Brisbane, CA) at ambient temperature in insulated packaging to minimize temperature fluctuation. The AlloSure test will be performed at the CareDx CLIA/CAP-accredited clinical laboratory. Samples will be tested, and results provided within 3 days of blood draw.
Diagnostic Test: AlloMap — AlloMap Kidney is intended to aid in the identification of SPK transplant recipients who have a low probability of rejection at the time in testing in conjunction with standard clinical assessment. For the AlloMap-Kidney test, approximately two tubes of blood will be obtained in PAXgene Blood RNA tubes and shipped to CareDx, Inc. (Brisbane, CA), where it will be tested.

SUMMARY:
This is a non-randomized, non-interventional, prospective pilot cohort study to monitor SPK patients post-transplant to determine if non-invasive measures using dd-cfDNA (Allosure) and AlloMap can assess an array of immune panels to predict and confirm the development of allograft injury and rejection in either organ.

Aims of the study

1. To develop and validate AlloSure and AlloMap in SPK transplant recipients with stable allograft function and in diagnosis of acute TCMR and ABMR in either organ
2. To assess the ability of AlloSure and AlloMap to determine early discordant rejection in SPK recipients
3. To investigate AlloSure and AlloMap in SPK transplant recipients with diagnosis of BKV viremia

DETAILED DESCRIPTION:
Currently, one the challenges of durable glucose management after pancreas transplantation is the ability to accurately and expediently diagnose early rejection to prevent unnecessary damage to the graft. This assessment is further complicated in combined organ transplantation. Simultaneous pancreas and kidney (SPK) transplantation accounts for most of the utilized pancreas grafts. However, both grafted systems (kidney and pancreas) are not subject to equal immunologic pressures even though they are theoretically presented with similar environments. Historically, the diagnosis of pancreatic rejection was assumed to be tethered to the presence of concomitant kidney rejection. The two organs were believed to reject in tandem. As such, many centers use sentinel biopsy of the kidney to determine rejection in the one or both organs. More recently, many studies have called into question this management strategy as there appears to be increasing evidence that both organs can reject independently of one another.

The presence of two organs allows for many combinations of rejection: both organs may undergo acute rejection known as concordant rejection or one organ may undergo acute rejection independently of the other organ known as discordant rejection. Kidney or pancreas rejection may occur in any time frame after SPK and can greatly affect graft survival. In order to clinically determine rejection in SPK recipients we monitor serum amylase, lipase, glucose, creatinine and proteinuria. Abnormalities in these labs in conjunction with clinical changes often are the indication for biopsy to determine the presence of rejection. More importantly, histology dictates treatment regimen and course. Invariably, SPK recipients sometimes present with normal creatinine and renal function, but with abnormal pancreatic enzymes. In most cases, the kidney biopsy would precede any discussion of pancreas biopsy due to the aforementioned notion of concordant rejection between organs. Certainly, biopsy proven rejection in the kidney with pancreatic enzymatic leak would necessitate aggressive anti-rejection therapy given the high likelihood of pancreatic involvement. However, many times these renal biopsies would be normal and lead to a quandary of how vigorously to pursue further evaluation of the pancreas.

Pancreas graft biopsy is not a common practice, but has been reported to be performed percutaneously, transcystoscopically if the pancreas was anastomosed to bladder, endoscopically, and laparoscopically in a few small series. Most centers use Interventional Radiology for CT guided pancreas biopsy. More importantly, there have been reported cases of complications for pancreas biopsies, mainly stemming from intraabdominal bleeding requiring surgical intervention [1]. In an effort to reduce potential patient morbidity from pancreatic biopsy, non-invasive tools like AlloSure that assesses donor-derived cell-free DNA (dd-cfDNA) and AlloMap; a gene expression-profiling test may provide an attractive alternative.

Currently dd-cfDNA analysis (AlloSure, CareDx®) in the kidney has shown promise. While the gold standard at present remains histologic assessment of kidney tissue, this may be changing as acceptance of dd-cfDNA grows. Dd-cfDNA analysis is advantageous as it is a noninvasive, less costly, and a potentially safer way to assess allograft rejection. Additionally, the easier accessibility of testing dd-cfDNA can enable more frequent testing, which can elucidate a more accurate progression of rejection rather than a biopsy which is only a snapshot in time. For renal analysis the recommended dd-cfDNA cutoff value is 1.0% to diagnose active rejection (positive and negative predictive values are 61% and 84%). While it seems reasonable that discordant rejection may apply to similar levels of dd-cfDNA seen in kidney alone rejection, concordant rejection levels of dd-cfDNA are unclear.

Notably, the technology behind Allosure has provided several insights into cellular injury from a variety of milieu. In the study by Shen et al., the dd-cfDNA level in deceased donors (44.99%) was significantly higher than that in the living donors (10.24%) at initial time, P < 0.01. Dd-cfDNA level in delayed graft function (DGF) recipients was lower (23.96%) than that in non-DGF (47.74%) at the initial time, P = 0.89 (19.34% in DGF and 4.46% in non-DGF on the first day, P = 0.17). There was a significant correlation between dd-cfDNA level at initial time and serum creatinine (r2 = 0.219, P = 0.032) and warm ischemia time (r2 = 0.204, P = 0.040). DGF patients experienced a slower decline than non-DGF patients, but both groups had a rapid decline in dd-cfDNA post-transplant.

However, most importantly it appears that a recurrence of dd-cfDNA level may be indicative of active rejection [5]. In the case report by Hurkmans et al., it was shown that dd-cfDNA was a sensitive biomarker to detect rejection in solid organ transplantation in a renal transplant patient diagnosed with melanoma and taking nivolumab as treatment. Additionally, the utility of Dd-cfDNA has been studied in the pediatric renal transplant population. In the study by Puliyanda et al., biopsies were completed when dd-cfDNA > 1.0% or when there was high clinical suspicion. 19 of 67 patients had dd-cfDNA testing as part of routine monitoring with a median dd-cfDNA score of 0.37 (IQR: 0.19-1.10). 48 of 67 patients who had clinical suspicion of rejection had median dd-cfDNA score of 0.47 (0.24-2.15). Donor specific antibody positive (DSA-positive) recipients had higher dd-cfDNA scores than those who were negative or had Angiotensin II Type 1 Receptor (AT1R) positivity alone (p = .003). There was no association between dd-cfDNA score and strength of DSA positivity. 7 of 48 recipients had a biopsy with a dd-cfDNA score <1%; two showed evidence of rejection. Neither DSA nor AT1R positivity was statistically associated with biopsy-proven rejection. However, dd-cfDNA >1% was diagnostic of rejection with sensitivity of 86% and specificity of 100% (AUC: 0.996, 0.98-1.00; P = .002). In the study by Sigdal et al., urinary dd-cfDNA after kidney transplantation correlates to the apoptotic injury load of the donor organ. Serial monitoring of urinary dd-cfDNA has been shown to be a sensitive proxy and biomarker of acute injury in the donor organ but fails to have specificity to differentiate between acute rejection and BK virus nephropathy. Therefore, dd-cfDNA is an appropriate and accurate method in lieu of a biopsy to assess allograft rejection and injury. However, one of the limitations of dd-cfDNA is its ability to be detected is inhibited by methylprednisolone.

In addition to donor-derived cell-free DNA (dd-cDNA), the quantification of select genes in circulating leukocytes (AlloMap, CareDx®) has potential to determine rejection. AlloMap has been shown to determine the risk for rejection in Cardiac Allograft Rejection Gene Expression Observational Trial (CARGO) and in the subsequent trial known as CARGO II. The current research of AlloMap in multi-organ recipients reflects a national cohort of 18 heart-kidney, 8 heart-liver, 1 heart-lung matched to 54 heart only recipients. AlloMap Heart® is a panel assay of 20 genes, 11 informative and 9 used for normalization and/or quality control, which produces gene expression data used in the calculation of an AlloMap Heart test score - an integer ranging from 0 to 40. Compared with patients in the same post-transplant period, the lower the score, the lower the probability of acute cellular rejection at the time of testing. Recently a multivariable gene-expression signature targeting T-cell-mediated rejection in peripheral blood of kidney transplant recipients was developed. This frugal TCMR-signature was made of (IFNG, IP-10, ITGA4, MARCH8, RORc, SEMA7A, WDR40A).

The gene expression profiles in renal transplant recipients with BKV viremia have been investigated by microarrays. This research analyzed entire blood gene expression profiles of 19 BKV viremia patients matched to 14 patients without BKV viremia and showed a significant higher expression of Gamma Interferon and Rejection-Induced Transcripts (GRIT), Cytotoxic T-cell-associated Transcripts (CAT), and Natural Killer cell-associated Transcripts (NK) cell associated transcript. The study results indicated increased activity of cytotoxic T cells and NK cells in both BKV viremia and nephropathy that resembled acute rejection and showed potential involvement of both the innate and adaptive immune system. This study documents to the importance of studying BKV viremia to exclude the diagnosis due to similar gene expression pattern in blood compared to rejection. In other study, gene expression profiles of DSA+ renal transplant recipients were analyzed with and without tissue findings of ABMR and found that DSA+ patients with ABMR has increased expression of activation, regulation, and differentiation of immune cells (T cells, NK cells, leukocytes, and interleukins).

Allosure and Allomap tests were not studied in SPK recipients in detail. Cutoff values for Allosure test could be different in stable SPK recipients compared to kidney transplant recipients due to additional donor tissue (pancreas and duodenum). It is also unknown, what would be the Allosure values in pancreas and/or kidney rejection in SPK recipients. It is also unknow the circulating gene transcripts in SPK recipients with rejection. Using the similar concept of peripheral blood gene expression by Allomap testing, AlloMap Kidney/Pancreas could be created.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study
* Male or Female, aged 18 years or above
* SKP transplant recipients between 1 month and 3 years after transplantation

Exclusion Criteria:

* Previous history of solid organ transplantation
* Pregnancy

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Simultaneous Pancreas-Kidney (SPK) transplant recipients will be enrolled at the time of transplantation or anytime within 3 years after transplantation starting at least 1 month after transplantation. Patients will have blood samples drawn at the time enrollment and at 3, 6, 9, and 12 months after enrollment and at the time of clinically indicated kidney and/or pancreas transplant biopsy. If the patients had biopsy proven acute or chronic rejection, Allosure and Allomap test will be repeated at 2, 4, and 6 weeks after the diagnosis. For patients who developed BKV viremia, Allosure and Allomap test will be tested at the time of BKV viremia and will be repeated at 2, 4, and 6 weeks after BKV viremia.
Sampling Method: Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2021-07-14 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Establishing benchmarks for AlloSure and AlloMap in SPK transplant recipients with stable allograft function | 3, 6, 9, and 12 months after enrolment
  Allosure score (%) and AlloMap test score (range 0-20) in stable kidney and pancreas transplant recipients

SECONDARY OUTCOMES:
To develop and validate AlloSure and AlloMap in SPK transplant recipients with diagnosis of acute TCMR and ABMR in either organ | 3, 6, 9, and 12 months after enrolment or at the time of clinically indicated kidney and/or pancreas biopsies and 2, 4, and 6 weeks after biopsy
  Allosure score (%) and AlloMap test score (range 0-20) in kidney and pancreas transplant recipients with rejection (TCMR or ABMR)

OTHER OUTCOMES:
AlloSure and AlloMap assessment in SPK transplant recipients with diagnosis of BKV viremia | 3, 6, 9, and 12 months after enrolment and at the time of BKV viremia and 2, 4 and 6 weeks after viremia
  Allosure score (%) and AlloMap test score (range 0-20) in kidney and pancreas transplant recipients with BKV viremia

CONTACTS AND LOCATIONS:
Overall Officials: Enver Akalin, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Klassen DK, Hoen-Saric EW, Weir MR, Papadimitriou JC, Drachenberg CB, Johnson L, Schweitzer EJ, Bartlett ST. Isolated pancreas rejection in combined kidney pancreas tranplantation. Transplantation. 1996 Mar 27;61(6):974-7. doi: 10.1097/00007890-199603270-00024. PMID 8623171
- [Background] Parajuli S, Arpali E, Astor BC, Djamali A, Aziz F, Redfield RR, Sollinger HW, Kaufman DB, Odorico J, Mandelbrot DA. Concurrent biopsies of both grafts in recipients of simultaneous pancreas and kidney demonstrate high rates of discordance for rejection as well as discordance in type of rejection - a retrospective study. Transpl Int. 2018 Jan;31(1):32-37. doi: 10.1111/tri.13007. Epub 2017 Aug 3. PMID 28672081
- [Background] Uva PD, Odorico JS, Giunippero A, Cabrera IC, Gallo A, Leon LR, Minue E, Toniolo F, Gonzalez I, Chuluyan E, Casadei DH. Laparoscopic Biopsies in Pancreas Transplantation. Am J Transplant. 2017 Aug;17(8):2173-2177. doi: 10.1111/ajt.14259. Epub 2017 Apr 4. PMID 28267898
- [Background] Bloom RD, Bromberg JS, Poggio ED, Bunnapradist S, Langone AJ, Sood P, Matas AJ, Mehta S, Mannon RB, Sharfuddin A, Fischbach B, Narayanan M, Jordan SC, Cohen D, Weir MR, Hiller D, Prasad P, Woodward RN, Grskovic M, Sninsky JJ, Yee JP, Brennan DC; Circulating Donor-Derived Cell-Free DNA in Blood for Diagnosing Active Rejection in Kidney Transplant Recipients (DART) Study Investigators. Cell-Free DNA and Active Rejection in Kidney Allografts. J Am Soc Nephrol. 2017 Jul;28(7):2221-2232. doi: 10.1681/ASN.2016091034. Epub 2017 Mar 9. PMID 28280140
- [Background] Shen J, Zhou Y, Chen Y, Li X, Lei W, Ge J, Peng W, Wu J, Liu G, Yang G, Shi H, Chen J, Jiang T, Wang R. Dynamics of early post-operative plasma ddcfDNA levels in kidney transplantation: a single-center pilot study. Transpl Int. 2019 Feb;32(2):184-192. doi: 10.1111/tri.13341. Epub 2018 Oct 2. PMID 30198148
- [Background] Hurkmans DP, Verhoeven JGHP, de Leur K, Boer K, Joosse A, Baan CC, von der Thusen JH, van Schaik RHN, Mathijssen RHJ, van der Veldt AAM, Hesselink DA. Donor-derived cell-free DNA detects kidney transplant rejection during nivolumab treatment. J Immunother Cancer. 2019 Jul 12;7(1):182. doi: 10.1186/s40425-019-0653-6. PMID 31300068
- [Background] Puliyanda DP, Swinford R, Pizzo H, Garrison J, De Golovine AM, Jordan SC. Donor-derived cell-free DNA (dd-cfDNA) for detection of allograft rejection in pediatric kidney transplants. Pediatr Transplant. 2021 Mar;25(2):e13850. doi: 10.1111/petr.13850. Epub 2020 Nov 20. PMID 33217125
- [Background] Sigdel TK, Vitalone MJ, Tran TQ, Dai H, Hsieh SC, Salvatierra O, Sarwal MM. A rapid noninvasive assay for the detection of renal transplant injury. Transplantation. 2013 Jul 15;96(1):97-101. doi: 10.1097/TP.0b013e318295ee5a. PMID 23756769
- [Background] Shen J, Guo L, Yan P, Zhou J, Zhou Q, Lei W, Liu H, Liu G, Lv J, Liu F, Huang H, Dong W, Shu L, Wang H, Wu J, Chen J, Wang R. Prognostic value of the donor-derived cell-free DNA assay in acute renal rejection therapy: A prospective cohort study. Clin Transplant. 2020 Oct;34(10):e14053. doi: 10.1111/ctr.14053. Epub 2020 Sep 4. PMID 32735352
- [Background] Deng MC, Eisen HJ, Mehra MR, Billingham M, Marboe CC, Berry G, Kobashigawa J, Johnson FL, Starling RC, Murali S, Pauly DF, Baron H, Wohlgemuth JG, Woodward RN, Klingler TM, Walther D, Lal PG, Rosenberg S, Hunt S; CARGO Investigators. Noninvasive discrimination of rejection in cardiac allograft recipients using gene expression profiling. Am J Transplant. 2006 Jan;6(1):150-60. doi: 10.1111/j.1600-6143.2005.01175.x. PMID 16433769
- [Background] Fujita B, Prashovikj E, Schulz U, Borgermann J, Sunavsky J, Fuchs U, Gummert J, Ensminger S. Predictive value of gene expression profiling for long-term survival after heart transplantation. Transpl Immunol. 2017 Mar;41:27-31. doi: 10.1016/j.trim.2017.02.001. Epub 2017 Feb 4. PMID 28167272
- [Background] Carey SA, Tecson KM, Jamil AK, Felius J, Wolf-Doty TK, Hall SA. Gene expression profiling scores in dual organ transplant patients are similar to those in heart-only recipients. Transpl Immunol. 2018 Aug;49:28-32. doi: 10.1016/j.trim.2018.03.003. Epub 2018 Mar 26. PMID 29588161
- [Background] Lubetzky M, Bao Y, O Broin P, Marfo K, Ajaimy M, Aljanabi A, de Boccardo G, Golden A, Akalin E. Genomics of BK viremia in kidney transplant recipients. Transplantation. 2014 Feb 27;97(4):451-6. doi: 10.1097/01.TP.0000437432.35227.3e. PMID 24310299
- [Background] Hayde N, Broin PO, Bao Y, de Boccardo G, Lubetzky M, Ajaimy M, Pullman J, Colovai A, Golden A, Akalin E. Increased intragraft rejection-associated gene transcripts in patients with donor-specific antibodies and normal biopsies. Kidney Int. 2014 Sep;86(3):600-9. doi: 10.1038/ki.2014.75. Epub 2014 Mar 26. PMID 24670411
- See also: Isolated pancreas rejection in combined kidney pancreas transplantation — https://pubmed.ncbi.nlm.nih.gov/8623171/
- See also: Concurrent biopsies of both grafts in recipients of simultaneous pancreas and kidney demonstrate high rates of discordance for rejection as well as discordance in type of rejection - a retrospective study — https://pubmed.ncbi.nlm.nih.gov/28672081/
- See also: Laparoscopic Biopsies in Pancreas Transplantation — https://pubmed.ncbi.nlm.nih.gov/28267898/
- See also: Cell-Free DNA and Active Rejection in Kidney Allografts — https://jasn.asnjournals.org/content/28/7/2221
- See also: Dynamics of early post-operative plasma ddcfDNA levels in kidney transplantation: a single-center pilot study — https://pubmed.ncbi.nlm.nih.gov/30198148/
- See also: Donor-derived cell-free DNA detects kidney transplant rejection during nivolumab treatment — https://jitc.biomedcentral.com/articles/10.1186/s40425-019-0653-6
- See also: A rapid noninvasive assay for the detection of renal transplant injury — https://pubmed.ncbi.nlm.nih.gov/23756769/
- See also: Prognostic value of the donor-derived cell-free DNA assay in acute renal rejection therapy: A prospective cohort study — https://pubmed.ncbi.nlm.nih.gov/32735352/
- See also: Noninvasive discrimination of rejection in cardiac allograft recipients using gene expression profiling — https://pubmed.ncbi.nlm.nih.gov/16433769/
- See also: Gene expression profiling scores in dual organ transplant patients are similar to those in heart-only recipients — https://pubmed.ncbi.nlm.nih.gov/29588161/
- See also: Genomics of BK viremia in kidney transplant recipients — https://pubmed.ncbi.nlm.nih.gov/24310299/